CLINICAL TRIAL: NCT05839119
Title: Targeting Androgen Signaling in Urothelial Cell Carcinoma - Neoadjuvant (TASUC-Neo): A Pilot Study of Degarelix in Combination With Neoadjuvant Gemcitabine and Cisplatin in Muscle-Invasive Urothelial Cell Carcinoma of the Bladder
Brief Title: Targeting Androgen Signaling in Urothelial Cell Carcinoma - Neoadjuvant
Acronym: TASUC-Neo
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: Legorreta Cancer Center at Brown University (Unknown); Lifespan (Other); Cures Within Reach (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BrUOG 428
Record Dates: First submitted 2023-04-20; First posted 2023-05-03 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Urothelial Carcinoma Bladder; Androgen Receptor Positive
Keywords: UCC; Bladder Cancer; AR+
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): In patients with androgen receptor positive (AR+), pT2 - pT4, N0 - N1, M0 urothelial cell carcinoma (UCC) of the bladder. The study medication, Degarelix, will be administered concurrently with neoadjuvant gemcitabine/cisplatin.
  * SOC Neoadjuvant Chemotherapy: Gemcitabine/Cisplatin 21-day cycles (4 cycles total)
  * Gemcitabine: 1000 mg/m2 (IV) Days 1 and 8 of each cycle
  * Cisplatin: 70 mg/m2 (if borderline renal function: 35 mg/m2) (IV) Day 1 of each cycle (if borderline renal function, days 1 and 8 of each cycle).
  * Study Medication: Degarelix (SC) Every 28-days (3 cycles total) Day -7 to -2 of cycle 1, then as defined in the study calendar (approximately q28 days). "initial dose is 240 mg administered as two 120 mg (3 mL) injections (SC), followed by subsequent doses at 80 mg (4 mL) administered as one injection (SC)
  Interventions: Drug: Degarelix; Combination Product: Gemcitabine/Cisplatin

INTERVENTIONS:
Drug: Degarelix — initial dose is 240 mg administered as two 120 mg (3 mL) injections (SC), followed by subsequent doses at 80 mg (4 mL) administered as one injection (SC)
  Other Names: Firmagon Kit
Combination Product: Gemcitabine/Cisplatin — SOC Neoadjuvant Chemotherapy: Gemcitabine/Cisplatin 21-day cycles (4 cycles total)
  * Gemcitabine: 1000 mg/m2 (IV) Days 1 and 8 of each cycle
  * Cisplatin: 70 mg/m2 (if borderline renal function: 35 mg/m2) (IV) Day 1 of each cycle (if borderline renal function, days 1 and 8 of each cycle).

SUMMARY:
This study is for patients who have bladder cancer that invades into the muscle wall of the bladder. The standard treatment for patients with muscle invasive bladder cancer is to give 4 cycles of chemotherapy with the drugs cisplatin and gemcitabine, then to do an operation to remove the bladder (cystectomy).

In this study, the investigators will test participants' bladder cancer to see if their bladder cancer has a receptor for testosterone inside the bladder cancer cells. If it has the testosterone receptor participants will receive a medication called Degarelix that lowers testosterone levels in the blood. Degarelix will be given during the period that participants are receiving the standard of care chemotherapy drugs gemcitabine and cisplatin.

The purpose of this study is to evaluate the effects, good and bad, of adding Degarelix to standard chemotherapy for patients with bladder cancer that have the testosterone receptor.

DETAILED DESCRIPTION:
Annually, over 80,000 people will be diagnosed with urothelial cell carcinoma (UCC) of the bladder in the USA, with over 17,000 deaths. For patients with muscle-invasive disease (stage II and IIIA), standard of care therapy is neoadjuvant chemotherapy followed by radical cystectomy. Neoadjuvant chemotherapy has been shown by multiple clinical trials and meta-analyses to improve pCR rates, disease free survival, and overall survival when compared to cystectomy alone. Specifically, neoadjuvant gemcitabine/cisplatin has been shown to be tolerable and effective and is a level 1 recommendation for treatment of muscle invasive bladder cancer by the National Comprehensive Cancer Network Guidelines.

The presence of a pCR in response to neoadjuvant chemotherapy is prognostic, but only about 35% of patients achieve a pCR. Thus improved neoadjuvant chemotherapy regimens are necessary to improve recurrence free survival and overall survival rates in patients with bladder cancer.

UCC is more common in men than women, with incidence rates of 3:1 to 4:1. This disparity persists even after controlling for smoking and occupational hazards/exposures and is likely influenced by androgen signaling. Androgen receptor (AR) positive UCC cells display increased proliferation, migration, and invasion in the presence of androgen and these effects are nullified in the presence of an AR antagonist. Preclinical studies show decreased rates of UCC incidence in response to a chemical carcinogen in castrated mice versus sham castrated mice and AR knockout mice versus AR intact mice. In retrospective human studies patients with UCC receiving androgen targeted therapy for concurrent prostate cancer had approximately 50% lower recurrence rates of UCC. Similarly, men receiving androgen targeted therapy for prostate cancer or benign prostatic hyperplasia have lower incidence rates of UCC than men not receiving androgen directed therapy.

Two prospective human clinical trials related to this concept have been performed. The first evaluated enzalutamide (an AR antagonist) as chemoprevention in non-muscle invasive UCC. This study was closed due to poor accrual after accruing only one patient. The second study added enzalutamide to standard chemotherapy in patients with metastatic UCC. Seven patients accrued at the therapeutic dose of enzalutamide. Overall, there was no signal for increased efficacy. However, one patient achieved a complete response lasting 2 years at last report. This patient was noted to have >90% positivity for AR in their tumor and, notably, was the only woman to participate in the study (and presumably had low testosterone levels). These data support further evaluation of androgen targeted therapy in AR+ UCC.

TASUC-neo is a pilot study conducted in patients with androgen receptor positive (AR+), pT2 - pT4, N0 - N1, M0 urothelial cell carcinoma (UCC) of the bladder. The study medication, Degarelix, will be administered concurrently with neoadjuvant gemcitabine/cisplatin.

ELIGIBILITY:
Inclusion Criteria:

3.1.1 Patients must have the following:

* Histologically confirmed muscle invasive urothelial cell carcinoma of the bladder (pT2 - pT4)
* Eligible for standard cisplatin/gemcitabine chemotherapy as determined by the treating Medical Oncologist

3.1.2 Patients must have muscle-invasive urothelial cell carcinoma of the bladder (pT2 - pT4, N0-N1, M0,) as determined by bladder biopsy or trans-urethral resection of bladder tumor (TURBT) and staging imaging studies. Patients with <10% non-urothelial histology will remain eligible for enrollment.

3.1.3 Androgen receptor positivity by IHC within the nucleus of tumor cells (as determined by study Pathologist) is required to receive study treatment.

3.1.4 Patients previously treated with intravesical therapy for non-muscle invasive urothelial carcinoma of the bladder are eligible for enrollment if the agent used was not gemcitabine or a platinum-containing agent (i.e, cisplatin, carboplatin, or oxaliplatin).

3.1.5 Age ≥18 years.

Because the safety and efficacy of Degarelix in pediatric patients have not been established, children (patients <18 years of age) are excluded from this study.

3.1.6 ECOG performance status ≤2 (Karnofsky ≥60%, see Appendix A).

3.1.7 Patients must have adequate organ and marrow function as defined below:

* absolute neutrophil count ≥1,000/mcL
* platelets ≥100,000/mcL
* total bilirubin ≤ institutional upper limit of normal (ULN)
* AST(SGOT)/ALT(SGPT) ≤3 1.5 × institutional ULN
* creatinine ≤ institutional ULN OR glomerular filtration rate (GFR) ≥40 mL/min/1.73 m2

3.1.8 Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.

3.1.9 For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.

3.1.10 Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.

3.1.11 Patients with metastases, including treated brain metastases, are not eligible for enrollment.

3.1.12 Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen, and prior therapy did not include gemcitabine or a platinum-containing agent, are eligible for this trial.

3.1.13 Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better.

3.1.14 For women of childbearing potential, a negative serum pregnancy test within 7 days prior to registration

3.1.15 Women of childbearing potential and male participants must practice highly effective form of non-hormonal contraception throughout the study, which is defined as from study screening (ICF) through at least six months post last treatment. It must be documented this was discussed with the patient.

The effects of Degarelix on the developing human fetus are unknown. However, based on animal studies and the mechanism of action, Degarelix may cause fetal loss. For this reason and that other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception.

3.1.16 Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

3.2.1 Patients who have previously received systemic or intravesical gemcitabine or platinum-containing chemotherapy

3.2.2 Patients taking testosterone, estrogen, or other sex hormone modifying agents are excluded from this study as these medications may interfere with the activity of the study drug, Degarelix.

3.2.3 Patients with uncontrolled intercurrent illness, as determined by the treating physician

3.2.4 Patients who are pregnant or breastfeeding. (The effects of Degarelix on the developing human fetus are unknown. However, "based on findings in animal studies, [Degarelix] can cause fetal harm and loss of pregnancy when administered to a pregnant woman. In animal developmental and reproductive toxicity studies in rats and rabbits, oral administration of Degarelix during organogenesis caused embryo-fetal lethality and abortion as well as increased post-implantation loss and decreased the number of live fetuses in animals at doses less than the clinical loading dose based on body surface area." (Degarelix package insert). For this reason and the fact that other therapeutic agents used in this trial are known to be teratogenic, pregnant women are excluded from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-10-02 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2032-01-01 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response rate (pCR) | Cystectomy following 4 (21-Day) cycles with Gemcitabine/Cisplatin
  Pathologic Complete Response (pCR): pCRis defined as no viable cancer cells in the resected bladder specimen.

SECONDARY OUTCOMES:
Rate of non-muscle invasive disease post neoadjuvant chemotherapy (ypT0, ypTis, ypTa, ypT1) | Cystectomy following 4 (21-Day) cycles with Gemcitabine/Cisplatin
  The effectiveness of the new combination will be assessed by pathological complete response rate (pCR). The exact one-sided 95% confidence intervals for the pCR will be reported.
Relapse free survival at 2 years | 2 yrs post Cystectomy
  Follow-up: from cystectomy. Year 1:q3 months, Year 2: q4 months
Relapse free survival at 5 years. | 5 yrs post Cystectomy
  Follow-up: Five years from cystectomy. Year 1:q3 months, Year 2: q4 months,Years 3: q6 months,Years 4: and 5: annually ( +\- 3-week window).
AR positivity in patients with a non-pCR at cystectomy | Cystectomy following 4 (21-Day) cycles with Gemcitabine/Cisplatin
  As a secondary analysis investigators will assess the rate of non-muscle-invasive disease and report the exact one-sided 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Sheldon L Holder, MD, PhD, Principal Investigator — Brown University
Locations (1):
- Lifespan Cancer Institute, Providence, Rhode Island, United States